CLINICAL TRIAL: NCT02157519
Title: Mobile Application for Improving Symptoms and Adherence to Oral Chemotherapy in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph A. Greer, Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-055
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-04

CONDITIONS: Adherence to Medication Regime; Cancer
Keywords: Oral Chemotherapy; Cancer
MeSH Terms: conditions — Medication Adherence; Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Application Intervention (Experimental): Participants in the intervention group will receive the mobile application for improving symptoms and adherence to oral chemotherapy along with their standard oncology care. The proposed elements of the mobile application include the following: 1) specification of an oral chemotherapy treatment plan; 2) weekly collection of patient-reported symptoms and medication adherence; and 3) delivery of real-time, tailored feedback to patients as well as immediate transmission of survey results to oncology clinicians.
  Interventions: Other: Mobile Application Intervention
- Standard Oncology Care (No Intervention): Participants in the control group will receive standard oncology care only.

INTERVENTIONS:
Other: Mobile Application Intervention — Participants assigned to the intervention group will receive the mobile application intervention for approximately three months after enrollment. The mobile app intervention will consist of completing an initial chemotherapy treatment plan, responding to weekly assessments regarding symptoms, side effects, and medication adherence, as well as receiving personalized feedback about responses. The results from patient surveys within the app will also be transmitted in real-time to the participants' oncology clinicians via a HIPAA-compliant, secure email.
  Arms: Mobile Application Intervention

SUMMARY:
Many people treated for cancer receive oral chemotherapy medications for their illness. This means that much of their cancer care occurs at home, away from a traditional oncology care setting. The purpose of this study is to explore how a Smartphone mobile application ("mobile app") can help improve the cancer treatment process in people who are prescribed oral chemotherapy medication. The investigators will explore how well the mobile app helps patients stay connected with their oncology care team, take their oral medications as prescribed, and manage their cancer-related symptoms from home. This study will be done in two phases: 1) a pilot phase to assess the feasibility of a mobile application intervention, and 2) a randomized-controlled trial to test the intervention.

DETAILED DESCRIPTION:
Background: Over the last decade, novel targeted agents have revolutionized the delivery of cancer care and improved survival rates, especially in those with metastatic disease. While oral chemotherapies possess significant advantages with respect to ease of administration, patients and caregivers receive less support for adherence and monitoring of side effects. Therefore, novel interventions are essential to help patients communicate in a more open and timely manner with their oncology clinicians to support adherence. As part of Phase 1 for this Patient-Centered Outcomes Research Institute (PCORI) grant, we conducted qualitative interviews with patients, clinicians and relevant stakeholders to inform the development of the proposed mobile app intervention. For the randomized-controlled trial, the investigators will recruit and randomly assign 180 adult patients prescribed oral chemotherapy to receive either the intervention (completed smartphone mobile app) or standard care.

Objective/Hypothesis: The goals of this study are to assess the feasibility and efficacy of a mobile application to help improve adherence to oral chemotherapy and symptom to patients with cancer. We will administer the intervention at three cancer centers, hypothesizing that patients with who use the mobile app will report better adherence to their oral chemotherapy and better management of symptoms than those patients who were not assigned to the intervention.

Specific Aims: The primary aims of this study are 1) to implement a patient-centered mobile application to assess symptoms, side effects, and adherence to oral chemotherapy that is feasible for use in oncology patients, and 2) to evaluate the efficacy of the mobile application in improving patient-reported clinical outcomes.

Study Design: We will recruit and randomly assign 180 patients from the three cancer care sites who have recently been prescribed oral chemotherapy to receive either the mobile app intervention or standard care. Participants will be stratified by study site (i.e. Massachusetts General Hospital (MGH), North Shore, MGH West, and Emerson Cancer Centers), cancer type, and line of chemotherapy. This will ensure relatively equal percentages of patients from each study site, diagnosis, and line of chemotherapy will be represented in the treatment and control groups. The mobile app intervention which will consist of completing an initial chemotherapy treatment plan with their oncology clinicians, responding to weekly assessments regarding symptoms, side effects, and medication adherence, as well as receiving personalized feedback about responses each week for 12 weeks. Medication adherence, symptom severity, and quality of life will serve as primary outcomes, and we will collect measures of quality cancer care as secondary targets. We will also explore whether particular patient characteristics (i.e. cancer type, demographics) affect patient response to the mobile app intervention.

ELIGIBILITY:
Inclusion Criteria:

Patient Participant Inclusion Criteria

* Age greater than 18 years
* Diagnosis of cancer with a new or existing prescription for oral chemotherapy
* Receiving cancer care at either Massachusetts General Hospital Cancer Center or community affiliates (North Shore or Emerson Hospitals)
* Eastern Cooperative Oncology Group (ECOG) ranging from 0 (asymptomatic) to 2 (symptomatic and in bed >50% of the day)
* Able to read and respond to questions in English
* Uses smart mobile phone (either operating system (iOS) [iPhone] or Android device)

Clinician Participant Inclusion Criteria - Clinician participants must be oncology clinicians (i.e. physicians and nurse practitioners) who maintain at least 25% clinical practice at the Massachusetts General Hospital Cancer Center or one of its community affiliates at the North Shore or Emerson Hospital.

Stakeholder Participant Inclusion Criteria - Four groups of stakeholders will provide ongoing feedback about the study design, methods, and results. To be eligible as a stakeholder, the participant must be able to represent the interests and perspective of at least one of the following stakeholder groups:

* Oncology Patient or Family Member
* Oncology Clinician (e.g., Physician or Nurse Practitioner)
* Cancer Practice Setting Administrator Health System, Community, and Society.

Exclusion Criteria:

Patient Participant Exclusion Criteria

* Individuals with co-morbid acute or untreated psychiatric symptoms (e.g., psychosis) or neurologic dysfunction will be excluded given that such symptoms would interfere with consent and participation.
* Individuals who own Windows or Blackberry smart mobile phones will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Greer, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital/North Shore Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital At Emerson Hospital-Bethke, Concord, Massachusetts

REFERENCES:
- [Derived] Fishbein JN, Nisotel LE, MacDonald JJ, Amoyal Pensak N, Jacobs JM, Flanagan C, Jethwani K, Greer JA. Mobile Application to Promote Adherence to Oral Chemotherapy and Symptom Management: A Protocol for Design and Development. JMIR Res Protoc. 2017 Apr 20;6(4):e62. doi: 10.2196/resprot.6198. PMID 28428158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2/13/15-12/31/16, patients with diverse malignancies were recruited from the outpatient oncology clinics at Massachusetts General Hospital Cancer Center and three community affiliates (i.e., Mass General/North Shore Cancer Center, Mass General Cancer Center at Mass General West, Mass General Cancer Center at Emerson Hospital-Bethke).
Pre-assignment Details: Of the 212 patients enrolled in our study, 181 were randomized. There were 28 participants who dropped out of the study after enrollment but prior to randomization, and 3 participants who were lost to follow-up after enrollment but prior to randomization.
Groups:
- Mobile Application Intervention: Mobile Application Intervention: Participants assigned to the intervention group received the mobile application intervention for approximately three months after enrollment. The mobile app intervention consisted of completing an initial chemotherapy treatment plan, responding to weekly assessments regarding symptoms, side effects, and medication adherence, as well as receiving personalized feedback about responses. The results from patient surveys within the app were transmitted weekly to the participants' oncology clinicians via a HIPAA-compliant, secure email.
- Standard Oncology Care: Participants in the control group received standard oncology care only, and completed baseline and post-assessments.
Period: Overall Study
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Started | 91 | 90
MEMScap Collected | 84 | 86
Completed | 80 | 89
Not Completed | 11 | 1
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Application Intervention | Standard Oncology Care | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13.7) | 53.8 (12.1) | 53.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 51 | 97
  Male | 45 | 39 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 87 | 82 | 169
  Unknown or Not Reported | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 84 | 75 | 159
  Asian | 6 | 4 | 10
  African American or Black | 0 | 5 | 5
  Hispanic/Latino/a | 0 | 4 | 4
  Multiracial | 0 | 2 | 2
  Other | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was collected from the Electronic Health Record based on oncologists' ratings.
  Scoring for the ECOG is as follows, with lower scores indicating a greater performance status:
  ECOG 0= Fully active, able to carry on all pre-disease performance without restriction ECOG 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work ECOG 2= Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    ECOG = 0 | 40 | 49 | 89
    ECOG = 1 | 47 | 40 | 87
    ECOG = 2 | 4 | 1 | 5
Cancer Type [Count of Participants; unit: Participants] — Type of cancer was collected from the Electronic Health Record
  Participants
    Hematologic | 30 | 30 | 60
    Non-small cell lung cancer | 17 | 16 | 33
    Breast | 11 | 15 | 26
    High grade Glioma | 9 | 12 | 21
    Sarcoma | 8 | 4 | 12
    Gastrointestinal | 6 | 2 | 8
    Melanoma | 4 | 3 | 7
    Genito-urinary | 4 | 3 | 7
    Low grade Glioma | 1 | 4 | 5
    Non-GIST Sarcoma | 1 | 1 | 2
Oral Therapy Type [Count of Participants; unit: Participants] — Type of prescribed oral therapy was collected from the Electronic Health Record.
  Participants
    Targeted therapy | 65 | 56 | 121
    Chemotherapy | 26 | 34 | 60

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Difficulties With Adherence on Any of the Four MMAS-4 Items in the Past Week
Description: The Morisky Medication Adherence Questionnaire (MMAS-4) - a 4-item questionnaire that assesses medication adherence in the past week by asking patients to indicate "yes" or "no" to each item (self-report). The four items ask patients to self-report whether they forgot to take their oral chemotherapy (OC) medication in the past week, whether they had any problems remembering to take their OC medication in the last week, whether they stopped taking their OC medication when they felt better in the past week, and whether they stopped taking their OC medication when they felt worse in the past week. Participants who answered "yes" to any of the four items were coded as having adherence problems, while those who indicated "no" to all four items were coded as having no adherence problems. Therefore, the count of participants is the number of participants who reported any difficulties with adherence on any of the four items in the past week.
Time Frame: Post-Assessment (12-14 weeks after baseline) controlling for baseline assessment
Population: Analysis population is the number of participants who completed the post-assessment measure of the MMAS-4
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Number analyzed (Participants) | 80 | 86
Participants | 11 | 20
Statistical Analysis 1: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the number of participants who self-reported adherence problems (i.e., dichotomous MMAS-4 scores) at post-assessment between groups adjusting for baseline self-reported adherence (i.e., dichotomous MMAS-4 scores) and change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.186, Regression, Logistic — threshold p <0.05; Adjusted for baseline MMAS-4 scores (dichotomous) and change in perceived social support (MSPSS) from baseline to post-assessment; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.23 to 1.33]

2. Primary Outcome: Adherence to Oral Chemotherapy Medication
Description: Medication Event Monitoring System (MEMS) utilizes an electronic pill cap to record the date and time the pill dispenser was opened.
Time Frame: Daily over course of study from baseline (within 2 weeks after enrollment) to post assessment (12-14 weeks after baseline)
Population: Analysis population is the number of participants who had data available from the Medication Event Monitoring System (MEMS) and completed the Multidimensional Scale of Perceived Social Support (MSPSS) at both the baseline and post assessments.
Measure: Mean (Standard Deviation); unit: percentage of medication taken
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Number analyzed (Participants) | 75 | 83
percentage of medication taken | 81.50 (2.93) | 79.16 (2.78)
Statistical Analysis 1: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the percentage of medication taken (as recorded by MEMS) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.57, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-10.35 to 5.68], Standard Error of Mean 4.06

3. Primary Outcome: Change in Symptoms and Side Effects
Description: M.D. Anderson Symptom Inventory (MDASI): a 19-item instrument that assesses the most common symptoms and side effects related to cancer and its treatment (self-report). The MDASI uses a 0-10 numerical rating scale for all items to assess the severity and interference of symptoms patients have experienced in the past 24 hours, with 0 being "not present" or "did not interfere" and 10 being "as bad as you can imagine" or "interfered completely". The ratings in the MDASI are averaged into two subscale scores: mean symptom severity (13 symptom items) and mean interference (6 interference items only), with possible scores on both subscales ranging from 0-10. Higher scores indicate worse symptom severity and interference, while lower scores indicate less symptom severity and interference.
Time Frame: Change score between 1) Baseline (within 2 weeks after enrollment) and 2) Post-Assessment (12-14 weeks after baseline)
Population: Participants who completed both baseline and post measures of the MDASI and the Multidimensional Scale of Perceived Social Support (MSPSS). Due to a clerical error, the MDASI was not administered to 31 pts at baseline. One pt skipped the symptom interference scale, causing a discrepancy in the number of pts completing each subscale on the MDASI.
Measure: Mean (Standard Error); unit: units on MDASI scale
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Number analyzed (Participants) | 67 | 71
units on MDASI scale
  Change in Symptom Severity | -0.03 (0.15) | 0.08 (0.15)
  Change in Symptom Interference: number analyzed (Participants) | 66 | 71
  Change in Symptom Interference | -0.12 (0.23) | -0.11 (0.23)
Statistical Analysis 1: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the change in symptom severity (MDASI-severity) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.603, Regression, Linear — threshold p <0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.31 to 0.53], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the change in symptom interference (MDASI-interference) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post assessment; Test type: Superiority; p = 0.982, Regression, Linear — threshold p <0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.64 to 0.65], Standard Error of Mean 0.33

4. Primary Outcome: Change in Quality of Life
Description: Functional Assessment of Cancer Treatment - General (FACT-G): a 27-item questionnaire that assesses physical, social, emotional, and functional well-being (self-report). The FACT-G utilizes a five-point scale from 0 (not at all) to 4 (very much). Four subscales are computed by taking the sum: physical well-being (7 items; range 0-28), social/family well-being (7 items; range 0-28), emotional well-being (7 items; range 0-24), and functional well-being (7 items; range 0-28). The overall score is the sum of the four subscale scores (range 0-108). Higher scores indicate greater quality of life, while lower scores indicate a worse quality of life.
Time Frame: Change score between 1) Baseline (within 2 weeks after enrollment) and 2) Post-Assessment (12-14 weeks after baseline)
Population: Analysis population is the number of participants who completed both baseline and post-assessment measures of the FACT-General (FACT-G) and the Multidimensional Scale of Perceived Social Support (MSPSS)
Measure: Mean (Standard Error); unit: units on the FACT-G scale
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Number analyzed (Participants) | 78 | 86
units on the FACT-G scale
  FACT-General: number analyzed (Participants) | 77 | 85
  FACT-General | 0.49 (1.19) | -1.93 (1.13)
  FACT-Physical Well-Being: number analyzed (Participants) | 77 | 86
  FACT-Physical Well-Being | 0.81 (0.48) | 0.11 (0.45)
  FACT-Social Well-Being | -0.55 (0.53) | -2.22 (0.50)
  FACT-Emotional Well-Being: number analyzed (Participants) | 78 | 85
  FACT-Emotional Well-Being | 0.04 (0.41) | 0.53 (0.40)
  FACT-Functional Well-Being | 0.35 (0.43) | -0.40 (0.41)
Statistical Analysis 1: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the change in overall QOL (FACT-G) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.144, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-5.66 to 0.83], Standard Error of Mean 1.65
Statistical Analysis 2: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the change in physical QOL (FACT-Physical Well-Being) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) baseline from baseline to post-assessment; Test type: Superiority; p = 0.294, Regression, Linear — threshold p <0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-2.00 to 0.61], Standard Error of Mean 0.66
Statistical Analysis 3: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the change in social QOL (FACT-Social Well-Being) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.025, Regression, Linear — threshold p <0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -1.67, 95% CI 2-sided [-3.12 to -0.21], Standard Error of Mean 0.74
Statistical Analysis 4: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the change in emotional QOL (FACT-Emotional Well-Being) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.392, Regression, Linear — threshold p <0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.64 to 1.63], Standard Error of Mean 0.58
Statistical Analysis 5: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the change in functional QOL (FACT-Functional Well-Being) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.216, Regression, Linear — threshold p <0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.94 to 0.44], Standard Error of Mean 0.60

5. Secondary Outcome: Treatment Satisfaction
Description: Description: Functional Assessment of Chronic Illness Treatment-Treatment Satisfaction-Patient Satisfaction (FACIT-TS-PS), 21-items that assesses patient satisfaction with doctor and staff competence, communication, and confidence and trust in providers, as well as overall satisfaction of care (self-report). The FACIT-TS-PS uses a 0-3 numerical rating scale to assess satisfaction with healthcare, with 0 representing the lowest level of satisfaction and 3 representing the highest level of satisfaction. Four subscales are computed by taking the sum: explanations (4 items; range 0-12), interpersonal (3 items, range 0-9), comprehensive care (7 items; range 0-21), nurses (3 items; range 0-9), and trust (4 items; range 0-12). A higher score indicates greater satisfaction with care, while a lower score represents lower satisfaction with care.
Time Frame: Change score between 1) Baseline (within 2 weeks after enrollment) and 2) Post-Assessment (12-14 weeks after baseline)
Population: Analysis population is the number of participants who completed both baseline and post-assessment measures of the FACIT-TS-PS and the Multidimensional Scale of Perceived Social Support (MSPSS)
Measure: Mean (Standard Deviation); unit: units on FACIT-TS-PS scale
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Number analyzed (Participants) | 78 | 86
units on FACIT-TS-PS scale
  FACIT-Clinician Explanations: number analyzed (Participants) | 78 | 85
  FACIT-Clinician Explanations | 0.04 (0.20) | -0.34 (0.19)
  FACIT-Interpersonal Treatment: number analyzed (Participants) | 78 | 84
  FACIT-Interpersonal Treatment | 0.07 (0.13) | -0.29 (0.13)
  FACIT-Comprehensive Care: number analyzed (Participants) | 77 | 85
  FACIT-Comprehensive Care | 0.08 (0.52) | -0.89 (0.49)
  FACIT-Nursing Care: number analyzed (Participants) | 77 | 82
  FACIT-Nursing Care | -0.45 (0.20) | -0.26 (0.19)
  FACIT-Trust in Clinicians: number analyzed (Participants) | 77 | 86
  FACIT-Trust in Clinicians | -0.24 (0.13) | -0.24 (0.12)
Statistical Analysis 1: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing change in treatment satisfaction with clinician explanations (FACIT-TS-PS-Clinician Explanations) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.170, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post assessment; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.93 to 0.17], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing change in satisfaction with interpersonal treatment (FACIT-TS-PS Interpersonal Treatment) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.057, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post assessment; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.72 to 0.01], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing change in treatment satisfaction with comprehensive care (FACIT-TS-PS Comprehensive Care) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.178, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-2.39 to 0.45], Standard Error of Mean 0.72
Statistical Analysis 4: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing change in treatment satisfaction with nursing care (FACIT-TS-PS Nursing Care) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.481, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.35 to 0.75], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing change in treatment satisfaction with trust in clinicians (FACIT-TS-PS Trust in Clinicians) from baseline to post-assessment between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.970, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.34 to 0.35], Standard Error of Mean 0.17

6. Secondary Outcome: Emergency Department Visits
Description: Resource Utilization Questionnaire, an adapted 3-item questionnaire inquiring about the number of emergency department visits and hospitalizations over the past three months (self-report). Patients are asked to indicate how many times they have gone to the emergency room in the past three months on a numerical scale ranging from 0 to "5 or more". Scores ranged from 0-5. A higher score represents more frequent emergency department visits, indicating higher resource utilization.
Time Frame: Post-Assessment (12-14 weeks after baseline)
Population: Analysis population is the number of participants who completed both baseline and post-assessment measures of the Resource Utilization Questionnaire (RUQ) and the Multidimensional Scale of Perceived Social Support (MSPSS)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Number analyzed (Participants) | 78 | 84
Scores on a scale | 0.16 (0.04) | 0.14 (0.04)
Statistical Analysis 1: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the number of emergency department (ED) visits over the study period between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.682, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.15 to 0.10], Standard Error of Mean 0.06

7. Secondary Outcome: Hospitalizations
Description: Description: Resource Utilization Questionnaire, an adapted 3-item questionnaire inquiring about the number of emergency department visits and hospitalizations over the past three months (self-report). Patients are asked to indicate how many times they have been admitted to the hospital in the past three months on a numerical scale ranging from 0 to "5 or more". Scores ranged from 0-5. A higher score represents more frequent hospital admissions, indicating higher resource utilization.
Time Frame: Post-Assessment (12-14 weeks after baseline)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mobile Application Intervention | Standard Oncology Care
Number analyzed (Participants) | 76 | 84
Scores on a scale | 0.20 (0.07) | 0.15 (0.07)
Statistical Analysis 1: Comparison: Mobile Application Intervention vs Standard Oncology Care; Analysis comparing the number of hospitalizations over they study period between groups adjusting for change in perceived social support (MSPSS) from baseline to post-assessment; Test type: Superiority; p = 0.640, Regression, Linear — threshold p < 0.05; Adjusted for change in perceived social support (MSPSS) from baseline to post-assessment; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.24 to 0.15], Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the active study period (study enrollment through post-assessment completion). As this was a behavioral intervention, adverse events were not assessed at any pre-specified time. Rather, they were recorded as reported by participants at any point during their study participation.
Description: As advanced cancer is a chronic-type illness, regular fluctuations in cancer-related symptoms, disease worsening, hospitalizations, emergency department visits, and deaths are to be expected, are not study-related, and will not be considered or reported as adverse events for the purposes of this study. Adverse events or unanticipated events that were study-related (e.g., security or privacy breaches) were reported to the IRB at the discretion of the PI.
Arm/Group | Mobile Application Intervention | Standard Oncology Care
All-Cause Mortality (participants affected / at risk) | 3/91 | 1/90
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/90
Other Adverse Events (participants affected / at risk) | 1/91 | 0/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobile Application Intervention (N=91) | Standard Oncology Care (N=90)
Adherence data of one study participant was lost in the mail (Product Issues) | 1 (1) | 0 (0) — A patient's de-identified Medication Event Monitoring System (MEMS) pill bottle was lost in the mail. There was no breach of confidentiality.

LIMITATIONS AND CAVEATS:
Due to a clerical error, the M.D. Anderson Symptom Inventory (MDASI) was not administered to 31 participants at baseline, which led to fewer cases available for analysis of change in this outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No